CLINICAL TRIAL: NCT03909711
Title: Relationship Between Temperature and Intraoperative Bleeding in Patients Undergoing Multilevel Spinal Surgery: Prospective, Multicenter Study
Brief Title: Relationship Between Temperature and Intraoperative Bleeding in Patients Undergoing Multilevel Spinal Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Federico Bilotta, Medical Doctor, Phisician Doctor, University of Roma La Sapienza
Other Study IDs: 5031
Record Dates: First submitted 2019-03-29; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Bleeding; Anemia
Keywords: Temperature; Bleeding; Anemia; Spine
MeSH Terms: conditions — Hemorrhage; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this multicentric observational study is to define the role of intraoperative temperature decrease (defined as reduction of at least 1 ° C during surgery) as haemorrhagic risk factor, evaluated as reduction of at least 1 gr / dl of hemoglobin, and to correlate it with the need for transfusion. Secondary objectives are infections and complications affecting other organs and systems incidence in the first week after surgery.

DETAILED DESCRIPTION:
In this prospective, observational, multicentric study, after ethics committee approval and patients informed consent, 20 patients for each center undergoing elective multi-level spine surgery procedures will be enrolled. A total of 80 patients will be enrolled. No randomization or concealment is planned.

Inclusion criteria are: adults (age> 18), American Society of Anesthesiologists (ASA) I-III, undergoing elective multi-level spinal surgery intervention. Patients with significant comorbidities such as severe liver disease, severe renal disease (stage III-IV), heart disease with organ failure, severe preoperative anemia requiring blood transfusions, severe pneumopathy with high probability of postoperative prolonged mechanical ventilation are excluded. Other exclusion criteria are: emergency intervention, known coagulopathy and chronic preoperative anemia.

Temperature will be measured with tympanic, anal or esophageal probe according to the availability and means of the department. Variables related to the patient (such as sex, age, BMI, smoke, anticoagulant or antiplatelet therapy in progress, presence of mild chronic hepatopathy / cardiopathy / pneumopathy / renal failure, hemoglobin and the preoperative hematocrit) will be compared with type and length of intervention, estimated blood loss, intraoperative variables (such as diuresis, minimum temperature and its variations, blood transfusions, ventilation mode) and post- operative hemoglobin level (the day after operation) to assess patient prognosis in terms of need for transfusion and infectious and respiratory complications incidence 7 days after surgery.

For each patient will be measured initial intraoperative temperature (T0) and minimum temperature (Tmin) with esophageal, anal or tympanic probe every 30 minutes during surgery. The temperature delta will be calculated as T0 - Tmin.

the investigators will compare intraoperative reduction of basal body temperature with Hb level reduction (preoperative Hb compared to Hb of the following day of intervention) considering as significant a temperature reduction of at least 1 ° C and Hb reduction of at least 1 g/dl, net of variables recognized correlated with increased bleeding in vertebral surgery (age, sex, diabetes mellitus, smoking, arterial hypertension, ASA class, intervention time, preoperative Ht) and liquid volume infused during intervention (hemodilution).

The continuous variables will be presented as mean and standard deviation while the categorical ones as frequency (percentage frequency, %).

Univariate logistic regression analysis will be applied to evaluate the effect of patients variables, surgical intervention with anesthesia management on patients prognosis in terms of need for transfusion and presence / absence of infectious and respiratory complications 7 days after surgery Variables associated with the need for transfusion and 7-day complications with p value <0.10 on univariate analysis will be considered in a multivariate logistic regression analysis model. The area under the receiver ROC curve (AUC) will be used as a measure of the model's prediction capacity.

ELIGIBILITY:
Inclusion Criteria:

* adults (age> 18)
* ASA I-III
* elective spinal surgery
* multi-level surgery

Exclusion Criteria:

* significant comorbidities such as severe liver disease, severe renal disease (stage III-IV), heart disease with organ failure, severe preoperative anemia requiring blood transfusions, severe pneumopathy with high probability of postoperative prolonged mechanical ventilation are excluded
* emergency intervention
* known coagulopathy
* chronic preoperative anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoig elective mulilevel spine surgery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
correlation between temperature and bleeding | the investigators are recruiting patients from November 2018 to November 2019
  the investigators aim to evaluate if temperature influence the bleeding of patients and which temperature seems to be the best (normothermia versus hypothermia). the investigators consider as significant bleeding the lost of at least 1 point of hemoglobin (lost >1mg/dl), and hypothermia the loss of at least 1°C of the body temperature

SECONDARY OUTCOMES:
Infections and complications related to bleeding | the investigators are recruiting patients from November 2018 to November 2019
  the investigators evaluate, with 1 week follow up, if there is any correlation between infections or other complications (pulmonary events, cardiac events...) and the bleeding of the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Policlinico Umberto I, University of Rome La Sapienza,, Rome, Italy